CLINICAL TRIAL: NCT04177979
Title: Efficacy of Near-Assisted Learning (NAL) in Improving Students' OSCE Grades: A Single-Blinded RCT
Brief Title: Efficacy of Near-Assisted Learning (NAL) in Improving Students' Objective Structured Clinical Examination (OSCE) Grades
Acronym: SRMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sulaiman AlRajhi Colleges (Other)
Responsible Party: Principal Investigator, Abdulaziz Alothman, Head of medical education department, Sulaiman AlRajhi Colleges
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SRMCOSCE
Record Dates: First submitted 2019-11-16; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Cost; Problem-based Learning; Peer Group
Keywords: Near-assisted learning; Cost; Education environment; OSCE; Problem-based learning

STUDY DESIGN:
Intervention Model Description: Randomized single blinded trial
Who Masked: Outcomes Assessor
Masking Description: The OSCE assessors were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near assisted learning group (Experimental): Participants in this arm were supervised by the trained peer-instructors.
  Interventions: Behavioral: Near-assisted learning through trained peers
- Self directed learning group (No Intervention): Participants in this arm were practicing independently. They were not supervised by any instructors.

INTERVENTIONS:
Behavioral: Near-assisted learning through trained peers — Students randomly allocated to this group were overseen during sessions by trained peer instructors.
  Arms: Near assisted learning group

SUMMARY:
This study aims to evaluate the impact of near-assisted learning (NAL) on first-year medical students' objective structured clinical examination (OSCE) grades in a problem-based learning (PBL) environment.

DETAILED DESCRIPTION:
In this randomized controlled trial, 1st year medical students were recruited in the study along with selected highly-performing, trained peer-instructors. The participants were randomly allocated to two groups, an intervention group supervised by the instructors and the control group that had to practice independently. They would attend OSCE sessions and had their performance evaluated, later on, in an exam. In addition to comparing their performance with each other, scores of the previous batch were considered in the comparison.

ELIGIBILITY:
Inclusion Criteria:

* 1st year medical students.
* Medical students of Sulaiman Alrajhi Colleges.
* Males.

Exclusion Criteria:

* Students of other academic levels.
* 1st year medical students of other universities.
* Females.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only males were recruited, due to sociocultural restrictions in Saudi Arabia
Enrollment: 48 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
objective structured clinical examination (OSCE) Score | Less than a month
  After the sessions, the study sample participated in the final osce exam. Their scores were compared. The minimum value was 0 while the maximum value was 100. The higher the score the better students had performed

CONTACTS AND LOCATIONS:
Locations (1):
- Sulaiman AlRajhi Colleges, Al Bukairiyah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Might be shared through the university webpage.

REFERENCES:
- [Result] Tolsgaard MG, Gustafsson A, Rasmussen MB, Hoiby P, Muller CG, Ringsted C. Student teachers can be as good as associate professors in teaching clinical skills. Med Teach. 2007 Sep;29(6):553-7. doi: 10.1080/01421590701682550. PMID 17978968
- [Result] Shah I, Mahboob U, Shah S. Effectiveness Of Horizontal Peer-Assisted Learning In Physical Examination Performance. J Ayub Med Coll Abbottabad. 2017 Oct-Dec;29(4):559-565. PMID 29330977
- [Result] Blank WA, Blankenfeld H, Vogelmann R, Linde K, Schneider A. Can near-peer medical students effectively teach a new curriculum in physical examination? BMC Med Educ. 2013 Dec 11;13:165. doi: 10.1186/1472-6920-13-165. PMID 24325639
- [Result] Riaz I. Peer assisted versus expert assisted learning: a comparison of effectiveness in terms of academic scores. J Coll Physicians Surg Pak. 2014 Nov;24(11):825-9. PMID 25404441
- [Result] Haist SA, Wilson JF, Brigham NL, Fosson SE, Blue AV. Comparing fourth-year medical students with faculty in the teaching of physical examination skills to first-year students. Acad Med. 1998 Feb;73(2):198-200. doi: 10.1097/00001888-199802000-00020. PMID 9484194
- [Result] Field M, Burke JM, McAllister D, Lloyd DM. Peer-assisted learning: a novel approach to clinical skills learning for medical students. Med Educ. 2007 Apr;41(4):411-8. doi: 10.1111/j.1365-2929.2007.02713.x. PMID 17430287
- [Result] Tai JH, Canny BJ, Haines TP, Molloy EK. The role of peer-assisted learning in building evaluative judgement: opportunities in clinical medical education. Adv Health Sci Educ Theory Pract. 2016 Aug;21(3):659-76. doi: 10.1007/s10459-015-9659-0. Epub 2015 Dec 12. PMID 26662035
- [Result] Liew SC, Sow CF, Sidhu J, Nadarajah VD. The near-peer tutoring programme: embracing the 'doctors-to-teach' philosophy--a comparison of the effects of participation between the senior and junior near-peer tutors. Med Educ Online. 2015 Sep 8;20:27959. doi: 10.3402/meo.v20.27959. eCollection 2015. PMID 26356229
- [Result] Tai J, Molloy E, Haines T, Canny B. Same-level peer-assisted learning in medical clinical placements: a narrative systematic review. Med Educ. 2016 Apr;50(4):469-84. doi: 10.1111/medu.12898. PMID 26995485
- [Result] Khaw C, Raw L. The outcomes and acceptability of near-peer teaching among medical students in clinical skills. Int J Med Educ. 2016 Jun 12;7:188-94. doi: 10.5116/ijme.5749.7b8b. PMID 27295403
- [Result] Cole JD, Ruble MJ, Donnelly J, Groves B. Peer-assisted Learning: Clinical Skills Training for Pharmacy Students. Am J Pharm Educ. 2018 Aug;82(6):6511. doi: 10.5688/ajpe6511. PMID 30181672
- [Result] Burke J, Fayaz S, Graham K, Matthew R, Field M. Peer-assisted learning in the acquisition of clinical skills: a supplementary approach to musculoskeletal system training. Med Teach. 2007 Sep;29(6):577-82. doi: 10.1080/01421590701469867. PMID 17978969
- [Result] Silbert BI, Lake FR. Peer-assisted learning in teaching clinical examination to junior medical students. Med Teach. 2012;34(5):392-7. doi: 10.3109/0142159X.2012.668240. Epub 2012 Apr 3. PMID 22471912
- See also: A non-pubmed indexed paper named: Improving Medical Student Confidence in Clinical Skills through a Peer-Facilitated Workshop — http://www.semanticscholar.org/paper/Improving-Medical-Student-Confidence-in-Clinical-a-Flynn-Williams/b5b6f1171bbd7c3e5d33ebb9644eb75aaaa5f8d1

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT04177979/Prot_SAP_000.pdf